CLINICAL TRIAL: NCT07195721
Title: The Effect of PROSE Treatment on Mental Health
Brief Title: The Effect of PROSE or Scleral Lenses on Mental Health
Status: Recruiting | Type: Observational
Sponsor: Boston Sight (Other)
Responsible Party: Sponsor
Other Study IDs: MH-2024-DB
Record Dates: First submitted 2025-09-25; First posted 2025-09-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-10

CONDITIONS: Depression - Major Depressive Disorder
Keywords: PROSE - prosthetic replacement of the ocular surface ecosystem

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who are considering PROSE treatment for ocular surface disease

SUMMARY:
The goal of this prospective clinical trial is to evaluate the effect that prosthetic replacement of the ocular surface ecosystem (PROSE, BostonSight, Needham MA) treatment may have on mental health, particularly affective mood disorders. Correlation between changes in mental health and ocular symptom improvement and/or visual function improvement will be evaluated.

DETAILED DESCRIPTION:
PROSE treatment is an FDA approved iterative process which includes designing a highly customized rigid gas permeable scleral lens for the treatment of ocular surface disease (such as keratoconjunctivitis sicca, Sjogren's syndrome, ocular Graft versus Host Disease and cicatricial keratoconjunctivitis) in order to mitigate pain (often severe), prevent vision loss from ocular surface breakdown, scarring, ulceration, melt and perforation and to achieve best corrected visual acuity. PROSE achieves its therapeutic purpose by filling the device each day with preservative free normal saline in order to neutralize corneal irregularities and to provide constant lubrication and protection to the ocular surface. Associations between mental health and ocular disease have been described in literature, including irregular corneas and ocular surface pathology. Many of these conditions are associated with dry eye symptoms. Given the role of inflammation in the pathogenesis of dry eye disease (DED) and the bidirectional nature of depression and inflammation, it is unsurprising that multiple studies have demonstrated the positive association between DED and anxiety and depression.

In particular, there is a strong association that those with depression may be more likely to have severe DED symptoms, with some studies showing increased likelihood of DED in patients with depression by an odds ratio of 1.92. Although the literature is inconsistent in its findings of the association between depression and objective DED signs, multiple studies have reliably shown that there is close alignment between subjectively reported DED symptoms and depression.

Mental health associations have also been established with ocular Graft versus Host Disease (oGvHD) both through the relationship between oGvHD and dry eye syndrome and as demonstrated by higher scores on Visual Function Questionnaire 25 (VFQ-25), which correlate to worse mental health status.

Patients with oGvHD report limitations in daily and recreational activities with some patients experiencing pain so severe that they are unable to leave their homes. Anecdotally, in clinical care, improvement with affect and mood are reported following treatment of these debilitating diseases with PROSE.

This is believed to be relatable to improvement in ocular symptoms, including pain, as well as improvement in vision and daily functionality.

This study will investigate the possible correlation of improved mental health following medical intervention with PROSE. The investigators hypothesize that patients with ocular surface disease who undergo first-time intervention with PROSE will demonstrate an improvement in mental health as measured by the validated PHQ-9 questionnaire19-23 within a 6-month timeframe. Investigators will also assess the relationship between changes in PHQ-9 scoring and ocular symptoms, utilizing the validated Ocular Surface Disease Index (OSDI). Lastly, investigators will evaluate the relationship between changes in PHQ-9 scoring and quality of life and functionality, utilizing the VFQ-25.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent has been obtained prior to any study-related procedures taking place.
2. Subject is Male or Female, 18 years of age or older prior to the initial visit.
3. Patient is proceeding with a PROSE or scleral lens consultation in one or both eyes for the primary diagnosis of ocular surface disease, including but not limited to Ocular Graft vs Host Disease, Keratoconjunctivitis Sicca, Dry eye, Sjogren's Disease, Rheumatologic ocular surface disease, Exposure Keratitis, Limbal Stem Cell Deficiency, Steven Johnson Syndrome, Mucous Membrane Pemphigoid (Ocular Cicatricial Pemphigoid), Atopic Keratoconjunctivitis, Chemical injury.
4. Baseline PHQ-9 score > 4
5. Baseline OSDI score of 13 or greater
6. In the opinion of the investigator, the subject can follow study instructions, complete all study procedures and visits
7. Is able to understand the English language in verbal and written interactions -

Exclusion Criteria:

1. Is currently participating in any other type of eye-related clinical research study that in the opinion of the investigator would interfere with the study
2. Is pregnant or nursing as reported by the subject.
3. Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study.
4. Recently started medication or other therapeutic treatments for affective mood disorders (such as depression) within the last 8 weeks.
5. Recently started new treatment for ocular surface disease, including but not limited to topical medicated drops, procedures, punctal plugs within the last 8 weeks.
6. Ocular surgery within the last 8 weeks
7. Planned ocular surgery within the study period
8. Has a known allergy to topical ophthalmic sodium fluorescein dye
9. Has a known intolerance to topical ophthalmic normal saline
10. Neurotrophic Keratitis
11. Corneal ectasia
12. PROSE or scleral lens wearer within the last 1 year prior to Visit 1 [subjects who have solely tried a PROSE or scleral lens in an office setting consultation (and were never dispensed for home use) ARE eligible for enrollment, regardless of whether it occurred in the last year]
13. Is an employee of BostonSight or an employee of a site performing the study -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are being evaluated for PROSE or scleral lens treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ9) | At enrollment, 28 days post PROSE dispense and 84 days post PROSE dispense
  The nine-item Patient Health Questionnaire (PHQ-9) is a depressive symptom scale and diagnostic tool introduced in 2001 to screen adult patients in primary care settings. The instrument assesses for the presence and severity of depressive symptoms and a possible depressive disorder. The minimum score on the PHQ9 is 0 and the maximum score is 27 which indicates the most severe depression.

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) questionnaire | At enrollment, 28 days post PROSE dispense and 84 days post PROSE dispense
  The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. The OSDI© is a valid and reliable instrument for measuring dry eye disease (normal, mild to moderate,and severe) and effect on vision-related function. The minimum score on the OSZDZI is 0 and the maximum score is 100 which indicates greater disability dues to dry eye disease.
Visual Function Questionnaire 25 (VFQ25) | At enrollment, 28 days post PROSE dispense and 84 days post PROSE dispense
  Measures the dimensions of self-reported vision-targeted health status that are most important for persons who have chronic eye diseases. The minimum score on the VFQ25 is 0 and the maximum score is 100 with higher scores indicating better visual function and health status.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Brocks, MD, Principal Investigator — Boston Sight
Locations (1):
- BostonSight, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided